CLINICAL TRIAL: NCT06220474
Title: Therapeutic Efficacy and Safety of Non-Invasive Radiofrequency Treatment in Patients With Refractory Meibomian Gland Dysfunction: A Randomized Controlled Trial
Brief Title: Therapeutic Efficacy and Safety of Non-Invasive RF Treatment in Refractory MGD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11221686
Record Dates: First submitted 2023-12-10; First posted 2024-01-24 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: One group of patients receiving radiofrequency treatment (RF) followed by meibomian gland expression (MGX) Another group of patients receiving and MGX
Who Masked: Participant, Investigator
Masking Description: It is a double-masked randomized study. Assigned treatment of a specific patients would be kept confidential in both the recruited participants and investigators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Radiofrequency treatment (RF), followed by meibomian gland expression (MGX) (Experimental): Before treatment, a thermage return pad will be applied to subject's skin to help prevent electrical burns. The return pad is a rubber, non-active electrode that creates a return path for radiofrequency energy back to the thermage comfort pulse technology (CPT) system. The upper and lower lid of both eyes are marked with skin marking paper (Thermage ® Skin Marking Paper TK-3.00). Coupling fluid is then applied to the external surface of the upper and lower lids of both eyes. All subjects then receive 225 applications to each eye over the upper and lower eyelids. Immediately after treatment, meibomian gland expression will be performed on both upper and lower eyelids of each eye for both eyes of all subjects using meibum expression forceps. Pain is minimized during this procedure by topical application of 0.4% oxybuprocaine hydrochloride.
  Interventions: Device: The Thermage FLX System
- Sham treatment, followed by meibomian gland expression (MGX) (Sham Comparator): The training mode is used in the Thermage FLX, which simulates treatment without dissipation of radiofrequency energy. Immediately after treatment, meibomian gland expression will be performed on both upper and lower eyelids of each eye for both eyes of all subjects using meibum expression forceps. Pain is minimized during this procedure by topical application of 0.4% oxybuprocaine hydrochloride.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: The Thermage FLX System — The Thermage FLX System is tested for its therapeutic efficacy and safety on treating refractory Meibomian Gland Dysfunction
  Arms: Radiofrequency treatment (RF), followed by meibomian gland expression (MGX)
Device: Sham treatment — Sham treatment acts as a control to test the therapeutic efficacy and safety of The Thermage FLX System
  Arms: Sham treatment, followed by meibomian gland expression (MGX)

SUMMARY:
The goal of this prospective, 24-week, double-masked, randomized, sham-controlled clinical trials to compare clinical efficacy and safety of RF and MGX with MGX alone in patients with meibomian gland dysfunction-related dry eye disease. The main question it aims to answer is whether radiofrequency treatment and meibomian gland expression is more effective in improving tear breakup time, as measured using non-invasive video keratography, compared with meibomian gland expression alone, in patients with refractory meibomian gland dysfunction-related dry eye disease.

Participants will be divided into two groups, one group will receive RF treatment followed with MGX and another will receive sham treatment with MGX.

DETAILED DESCRIPTION:
Dry eye disease(DED) is a prevalent age-related ophthalmic condition. Depending on the population studied and the diagnostic criteria used, dry eye disease is estimated to have a high prevalence in most populations , with a female preponderance. In the latest 2017 Tear Film and Ocular Surface Society Dry Eye Workshop II (TFOS DEWS II) Epidemiology Report, which compiled dry eye prevalence data from studies worldwide, the reported the prevalence of DED ranged from 5 to 50%. The risk of dry eye disease increases with age, where with every increase in 10 years of age, the self-reported symptoms of DED increased by 2%. In one study in Asia, up to 70% of elderly patients greater than 60 years of age suffering from symptomatic dry eye disease. Dry eye disease causes gritty and painful eyes, with associated blurred vision. For sufferers, it poses a significant burden on quality of life and limitations activities on activities of daily living, resulting in considerable economic costs to society. A 2006 health-economics study in the United Kingdom estimated that the annual healthcare costs to the public sector for every 1000 dry eye patients was USD 1.1 million.

The causes of dry eye can be broadly classified into those with aqueous tear deficiency, excessive tear evaporation or a combination of both. The most common cause of excessive tear evaporation is meibomian gland dysfunction (MGD). This is a common condition of the eyelids where there is a significant change in both the consistency and quantity of meibum, resulting in chronic inflammation of the eyelids and subsequent ocular surface dysfunction. MGD has a prevalence from 46.2% to 69.3% in several studies targeting Asian populations, with a trend of higher prevalence in the elderly. Insufficient lipid secretion from meibomian gland undermines tear film stability, producing dry eye symptoms despite normal tear secretion. In a recent study, up to 70.3% of dry eye patients were found to have concurrent MGD. Refractory MGD is defined by the failure to respond to more than at least three types of conventional therapy, including lubricating eyedrops, gels and ointments and topical or systemic anti-inflammatory treatment, in the past two years.

Currently heat-based therapies are the mainstay and most effective strategies against MGD. Eyelid warming, thermal pulsation and intense light therapy are three prevailing heat-based treatments for MGD- related dry eye disease. Eyelid warming usually involves the application of warm towels, commercialized eye masks (EyeGiene® or Blephasteam®) or eye bags (MGDRx Eye Bag) at least twice a day. Thermal pulsation (Lipiflow®) refers to the delivery of controlled heat together with gentle massage to the eyelids by the machine for 10-17 minutes. Intense pulsed light (IPL) therapy, which uses light energy on the skin surface, is widely used in dermatology to treat a variety of conditions including dermal vascular lesions, such as port wine stains and hemangiomas, facial rosacea, and acne. Each treatment strategy however carries significant limitations. Self-applied eyelid warm compress is cheap and easily available, but when used alone has limited efficacy. Furthermore, sustained patient adherence to treatment is difficult long term. A single treatment of thermal pulsation therapy has been shown to have sustained therapeutic effects up to 12 months after treatment. However, thermal pulsation is not effective in moderate to severe cases of MGD. From existing studies, IPL has greater clinical efficacy than thermal pulsation, but its therapeutic effects are maintained for a significantly shorter period. As such, monthly repeated treatments for up to 8 months may be required for sustained effects. It is also important to note that none of the existing treatments allow the eyelids to evacuate inspissated meibum effectively, with meibum expression by an ophthalmologist an important step in the treatment process. Thus, MGD is likely to recur long-term.

The Thermage FLX System (WA, USA) is a non-ablative radiofrequency (RF) energy-based device, which has been widely adopted in the cosmetic industry for radiofrequency tissue tightening. RF transfers high energy fluences through the skin to deep dermal layers uniformly while protecting the epidermis. It is postulated that RF stimulates subdermal collagen production for tissue tightening effect. There are several advantages of using non-invasive RF treatment over other currently available energy-based devices. Firstly, the Thermage FLX has a much more precise applicator directly targeting the meibomian glands. Thermage FLX addresses both the upper and lower eyelids as close as possible to the lid margin, which is directly where the meibomian glands are situated, it also addresses the tragus area as well, hence a more precise and direct treatment area can be achieved. Secondly, compared to other energy-based devices, Thermage FLX provides a higher accumulative heat transfer effect around the periocular region, due to its repeated application of at least 4-5 cycles around the periorbital region. With higher accumulative heat energy, we anticipate a better and more effective melting of the meibum, which aids in more effective meibum expression. Thirdly, as Thermage FLX has been widely adopted for radiofrequency tissue tightening due to its collagen resynthesis effect, there has been proven improvement of the elasticity of orbicularis and periocular skin tissue, this can promote better blinking effort and better apposition of lid margins. This may enhance the pumping effect of the orbicularis oculi in the long-term. RF treatment is potentially a safe and effective multimodal treatment for MGD-related dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or more
2. Bilateral dry eye disease as confirmed by presence of both symptoms and signs 2.1 Symptoms: Abnormal result on the Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) dry eye symptom questionnaire (≥5) 2.2 Signs: Abnormal result in at least one of the following three clinical tests - tear osmolarity, NIKBUT and corneal staining for punctate epithelial erosions and,
3. Bilateral moderate to severe meibomian gland dysfunction - at least Grade 1 meibum quality (cloudy appearance) and Grade 2 meibum expressibility (moderate pressure required). And,
4. Refractory MGD - The failure to respond to at least three types of conventional therapy, including artificial tears, topical or systemic antibiotics and anti-inflammatory treatments and the aforementioned heat-based therapies, over a period of at least 2 years
5. Fitzpatrick skin type I-IV - Type V and VI skinned subjects are excluded from the study due to the high risk of pain and focal hypopigmentation
6. Mentally fit to give informed consent

Exclusion Criteria:

1. Fitzpatrick skin type V-VI
2. History of eyelid scarring
3. Infrared meibography evidence of significant acinar gland atrophy (dropout of >30%) - these patients have been shown not to benefit from heat-based therapies due to end-stage disease
4. Pregnancy or lactation
5. Active corneal disease such as infectious keratitis, allergic keratoconjunctivitis, pterygium, exposure keratopathy, lagophthalmos, trichiasis or dellen
6. Current systemic intake of photosensitive medications, including tetracycline group of drugs.
7. History of corneal abnormality or surgery within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in non-invasive keratographic tear breakup time (NIKBUT) | From baseline to 6 months post- treatment between study groups
  NIKBUT is measured in seconds and average of 3 consecutive readings is taken. Higher values mean better outcomes.

SECONDARY OUTCOMES:
Change in Standard Patient Evaluation of Eye Dryness (SPEED) symptom score | From baseline to 6 months post-treatment between study groups
  One number was collected per patient, with higher scores meaning worse outcomes
Percentage of subjects with normal non-invasive keratographic tear breakup time (NIKBUT) | 6 months
  > 10 seconds, with lower scores meaning worse
Percentage of subjects with normal SPEED | 6 months
  <5, with higher scores meaning worse
Change in best corrected visual acuity | from baseline to 6 months post-treatment
  from logmar(1.0 to -0.1)
Incidence of periorbital pain | 6 months
  at least 3/10 and above, with higher scores meaning worse
Incidence of ocular adverse events | 6 months
  evidence of uveitis, conjunctivitis, scleritis/episcleritis, new lens opacities, new cornea opacities
Incidence of non-ocular adverse events | 6 months
  eyelid skin burn, eyelid redness, eyelid hyper/hypopigmentation

OTHER OUTCOMES:
Change in cornea staining (National Eye Institute Grading System) | from baseline to 6 months post-treatment
  This serves as an objective parameter for ocular surface damage, with higher scores meaning worse
Tear osmolarity | from baseline to 6 months post-treatment
  This serves as an objective parameter for ocular surface damage
Change in Shirmer's I test reading | from baseline to 6 months post-treatment
  In millimetres. Readings serve as objective parameters for tear volume
Tear meniscus height | from baseline to 6 months post-treatment
  In millimetres. Readings serve as objective parameters for tear volume
Changes in meiboscore | from baseline to 6 months post-treatment between study groups
  These readings serve as parameters for meibomian gland dysfunction
Changes in meibum expressibility | from baseline to 6 months post-treatment between study groups
  These readings serve as parameters for meibomian gland dysfunction, with higher scores meaning worse
Changes in meibum quality | from baseline to 6 months post-treatment between study groups
  These readings serve as parameters for meibomian gland dysfunction, with higher scores meaning worse

CONTACTS AND LOCATIONS:
Overall Officials: Kendrick Co SHIH, Principal Investigator — The University of Hong Kong, Grantham Hospital
Locations (2):
- Hong Kong (2):
  - Grantham Hospital, Hong Kong
  - HKU Eye Centre, Hong Kong

REFERENCES:
- [Background] McCarty CA, Bansal AK, Livingston PM, Stanislavsky YL, Taylor HR. The epidemiology of dry eye in Melbourne, Australia. Ophthalmology. 1998 Jun;105(6):1114-9. doi: 10.1016/S0161-6420(98)96016-X. PMID 9627665
- [Background] Lee AJ, Lee J, Saw SM, Gazzard G, Koh D, Widjaja D, Tan DT. Prevalence and risk factors associated with dry eye symptoms: a population based study in Indonesia. Br J Ophthalmol. 2002 Dec;86(12):1347-51. doi: 10.1136/bjo.86.12.1347. PMID 12446361
- [Background] Chia EM, Mitchell P, Rochtchina E, Lee AJ, Maroun R, Wang JJ. Prevalence and associations of dry eye syndrome in an older population: the Blue Mountains Eye Study. Clin Exp Ophthalmol. 2003 Jun;31(3):229-32. doi: 10.1046/j.1442-9071.2003.00634.x. PMID 12786773
- [Background] Lin PY, Tsai SY, Cheng CY, Liu JH, Chou P, Hsu WM. Prevalence of dry eye among an elderly Chinese population in Taiwan: the Shihpai Eye Study. Ophthalmology. 2003 Jun;110(6):1096-101. doi: 10.1016/S0161-6420(03)00262-8. PMID 12799232
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Moss SE, Klein R, Klein BE. Prevalence of and risk factors for dry eye syndrome. Arch Ophthalmol. 2000 Sep;118(9):1264-8. doi: 10.1001/archopht.118.9.1264. PMID 10980773
- [Background] Stapleton F, Alves M, Bunya VY, Jalbert I, Lekhanont K, Malet F, Na KS, Schaumberg D, Uchino M, Vehof J, Viso E, Vitale S, Jones L. TFOS DEWS II Epidemiology Report. Ocul Surf. 2017 Jul;15(3):334-365. doi: 10.1016/j.jtos.2017.05.003. Epub 2017 Jul 20. PMID 28736337
- [Background] Mathers WD, Lane JA, Zimmerman MB. Tear film changes associated with normal aging. Cornea. 1996 May;15(3):229-34. doi: 10.1097/00003226-199605000-00001. PMID 8713923
- [Background] Moss SE, Klein R, Klein BE. Incidence of dry eye in an older population. Arch Ophthalmol. 2004 Mar;122(3):369-73. doi: 10.1001/archopht.122.3.369. PMID 15006852
- [Background] The epidemiology of dry eye disease: report of the Epidemiology Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):93-107. doi: 10.1016/s1542-0124(12)70082-4. PMID 17508117
- [Background] Miljanovic B, Dana R, Sullivan DA, Schaumberg DA. Impact of dry eye syndrome on vision-related quality of life. Am J Ophthalmol. 2007 Mar;143(3):409-15. doi: 10.1016/j.ajo.2006.11.060. Epub 2007 Jan 2. PMID 17317388
- [Background] Clegg JP, Guest JF, Lehman A, Smith AF. The annual cost of dry eye syndrome in France, Germany, Italy, Spain, Sweden and the United Kingdom among patients managed by ophthalmologists. Ophthalmic Epidemiol. 2006 Aug;13(4):263-74. doi: 10.1080/09286580600801044. PMID 16877285
- [Background] Foulks GN, Bron AJ. Meibomian gland dysfunction: a clinical scheme for description, diagnosis, classification, and grading. Ocul Surf. 2003 Jul;1(3):107-26. doi: 10.1016/s1542-0124(12)70139-8. PMID 17075643
- [Background] Schaumberg DA, Nichols JJ, Papas EB, Tong L, Uchino M, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on the epidemiology of, and associated risk factors for, MGD. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1994-2005. doi: 10.1167/iovs.10-6997e. Print 2011 Mar. No abstract available. PMID 21450917
- [Background] Rabensteiner DF, Aminfar H, Boldin I, Schwantzer G, Horwath-Winter J. The prevalence of meibomian gland dysfunction, tear film and ocular surface parameters in an Austrian dry eye clinic population. Acta Ophthalmol. 2018 Sep;96(6):e707-e711. doi: 10.1111/aos.13732. Epub 2018 Apr 15. PMID 29656524
- [Background] Lam PY, Shih KC, Fong PY, Chan TCY, Ng AL, Jhanji V, Tong L. A Review on Evidence-Based Treatments for Meibomian Gland Dysfunction. Eye Contact Lens. 2020 Jan;46(1):3-16. doi: 10.1097/ICL.0000000000000680. PMID 31834043
- [Background] Toyos R, McGill W, Briscoe D. Intense pulsed light treatment for dry eye disease due to meibomian gland dysfunction; a 3-year retrospective study. Photomed Laser Surg. 2015 Jan;33(1):41-6. doi: 10.1089/pho.2014.3819. PMID 25594770
- [Background] Wang MT, Jaitley Z, Lord SM, Craig JP. Comparison of Self-applied Heat Therapy for Meibomian Gland Dysfunction. Optom Vis Sci. 2015 Sep;92(9):e321-6. doi: 10.1097/OPX.0000000000000601. PMID 25955642
- [Background] Gupta PK, Vora GK, Matossian C, Kim M, Stinnett S. Outcomes of intense pulsed light therapy for treatment of evaporative dry eye disease. Can J Ophthalmol. 2016 Aug;51(4):249-253. doi: 10.1016/j.jcjo.2016.01.005. Epub 2016 Jun 22. PMID 27521662
- [Background] Vegunta S, Patel D, Shen JF. Combination Therapy of Intense Pulsed Light Therapy and Meibomian Gland Expression (IPL/MGX) Can Improve Dry Eye Symptoms and Meibomian Gland Function in Patients With Refractory Dry Eye: A Retrospective Analysis. Cornea. 2016 Mar;35(3):318-22. doi: 10.1097/ICO.0000000000000735. PMID 26785301
- [Background] Hodgkinson DJ. Clinical applications of radiofrequency: nonsurgical skin tightening (thermage). Clin Plast Surg. 2009 Apr;36(2):261-8, viii. doi: 10.1016/j.cps.2008.11.006. PMID 19309652
- [Background] Sukal SA, Geronemus RG. Thermage: the nonablative radiofrequency for rejuvenation. Clin Dermatol. 2008 Nov-Dec;26(6):602-7. doi: 10.1016/j.clindermatol.2007.09.007. PMID 18940540
- [Background] Fitzpatrick R, Geronemus R, Goldberg D, Kaminer M, Kilmer S, Ruiz-Esparza J. Multicenter study of noninvasive radiofrequency for periorbital tissue tightening. Lasers Surg Med. 2003;33(4):232-42. doi: 10.1002/lsm.10225. PMID 14571447